CLINICAL TRIAL: NCT05852119
Title: Prospective Study for the Outpatient Treatment of Patients With Very Low Risk Acute Symptomatic Pulmonary Embolism. TRAMTEP Study.
Brief Title: Prospective Study for the Outpatient Treatment of Patients With Very Low Risk Acute Symptomatic Pulmonary Embolism.
Acronym: TRAMTEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 295-22
Record Dates: First submitted 2023-04-26; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-04

CONDITIONS: Acute Pulmonary Embolism; Outpatient Treatment
MeSH Terms: interventions — Ambulatory Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemodynamically stable patients with very low risk symptomatic acute pulmonary embolism (PE) (Experimental)
  Interventions: Other: Outpatient treatment with standard anticoagulant therapy

INTERVENTIONS:
Other: Outpatient treatment with standard anticoagulant therapy — All patients included in the study will be treated on an outpatient basis, that is, they will be discharged within the first 24 hours of the diagnosis of PE in the Emergency Department.

SUMMARY:
Objectives: To evaluate the safety of outpatient treatment of patients with very low-risk pulmonary embolism (PE), and the satisfaction and quality of life of this management.

Methods: An experimental study of routine clinical practice will be carried out in which 300 consecutive hemodynamically stable patients with acute symptomatic PE will be included, who meet all the inclusion criteria and none of the exclusion criteria. All patients included in the study will be treated on an outpatient basis, that is, they will be discharged within the first 24 hours of the diagnosis of PE in the Emergency Department. The Computerized Registry of Thromboembolic Disease RIETE (Registro Informatizado de Enfermedad TromboEmbólica) will be used to collect the data in electronic case report form (CRF) and ensure the quality of the data.

Setting: Emergency, Pneumology and Internal Medicine Services of 10 Spanish hospitals.

Analysis: An intention-to-treat (ITT) analysis will be performed on all patients who sign the informed consent and are included in the study (regardless of whether or not they receive the assigned strategy). Additionally, an analysis of all patients who are treated on an outpatient basis without deviations or violations of the protocol will be performed. The primary outcome considered will be the composite of recurrent PE, major bleeding, or death from any cause during the first 30 days after enrollment in the study. Patient satisfaction and quality of life will be considered as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of suspected pulmonary embolism (PE) by multidetector chest angio computed tomography (CT), if a contrast-encircled partial intraluminal defect or complete pulmonary artery occlusion is demonstrated on two consecutive CT slices (13);
* Right ventricle (RV) diameter equal to or less than that of the left ventricle (LV) (RV/LV ratio ≤1) on chest CT angiography (see Study Procedures); and
* Negatively modified simplified Pulmonary Embolism Severity Index (sPESI) scale at the time of evaluation of the patient in the Emergency Department.

Exclusion Criteria:

* Inability to obtain informed consent
* Pregnancy
* Hemodynamic instability at diagnosis (defined by systolic blood pressure (SBP) <90 mm Hg, indication of fibrinolytic treatment or inferior vena cava filter, need for vasoactive drugs at the discretion of the attending physician, cardiopulmonary resuscitation or orotracheal intubation)
* Contraindication for anticoagulation, at the discretion of the responsible physician;
* Estimated survival of less than 3 months
* Need for thrombectomy, vena cava filter insertion, or need for fibrinolytic treatment of the PE episode at the time of diagnosis
* Participation in a clinical trial for the treatment of venous thromboembolic disease
* Impossibility of follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Composite of recurrent pulmonary embolism (PE), major bleeding, or death from any cause. | 30 days
  The primary outcome considered will be the composite of recurrent PE, major bleeding, or death from any cause during the first 30 days after enrollment in the study.

SECONDARY OUTCOMES:
Satisfaction of the patients | 30 days
  The satisfaction of the patients will be evaluated on day 30 of follow-up using the Patient Satisfaction Questionnaire (PSQ-18).
Quality of life of the patients | 30 days
  Quality of life of the patients will be evaluated on day 30 of follow-up using the Pulmonary Thromboembolism Quality of Life Questionnaire (PEmb-Qol).

CONTACTS AND LOCATIONS:
Overall Officials: PEDRO Ruiz-Artacho, PhD, MD, Study Director — Clínica Universidad de Navarra, Madrid (España); Raquel Morillo Guerrero, PhD, MD, Study Director — Hospital Ramón y Cajal, Madrid (España); DAVID Jiménez Castro, PhD, MD, Study Director — Hospital Ramón y Cajal, Madrid (España); Deisy Barrios Barreto, PhD, MD, Study Director — Hospital Ramón y Cajal, Madrid (España); Pablo Demelo Rodríguez, PhD, MD, Principal Investigator — Hospital Universitario Gregorio Marañón, Madrid (España); Alberto García-Ortega, PhD, MD, Principal Investigator — Hospital Doctor Peset, Valencia (España); Andrea Pérez Figuera, MD, Study Director — Hospital Ramón y Cajal, Madrid (España); Elena Hernando López, MD, Principal Investigator — Hospital San Pedro, Logroño (España); Luis Jara Palomares, PhD, MD, Principal Investigator — Complejo Hospitalario Virgen del Rocío, Sevilla (España); Jorge Moisés Lafuente, MD, Principal Investigator — Hospital Clinic (España); Ignacio Casado Moreno, MD, Principal Investigator — Hospital Universitario Virgen de las Nieves, Granada (España; Tina Rivas, MD, Principal Investigator — Hospital Universitario Donostia (España); Daniel Segura Ayala, MD, Principal Investigator — Hospital General Universitari de Castelló (España)
Locations (10):
- Spain (10):
  - Hospital Clinic, Barcelona
  - Hospital General Universitari de Castelló, Castelló
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital San Pedro, Logroño
  - Clínica Universidad Navarra, Madrid
  - Hospital Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Complejo Hospitalario Virgen del Rocío, Seville
  - Hospital Doctor Peset, Valencia